CLINICAL TRIAL: NCT06766084
Title: Is Total Arterial Revascularization Superior to Multiarterial Grafting in Coronary Artery Bypass Grafting
Status: Completed | Type: Observational
Sponsor: Technion, Israel Institute of Technology (Other)
Responsible Party: Principal Investigator, Dror B. Leviner, Director of advanced cardiac surgery Department of cardiac surgery Carmel medical center, Technion, Israel Institute of Technology
Other Study IDs: RMC - 22-169
Record Dates: First submitted 2025-01-02; First posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: CABG; Revascularization

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- multiarterial grafting
  Interventions: Procedure: CABG
- total arterial revascularization
  Interventions: Procedure: CABG

INTERVENTIONS:
Procedure: CABG — All patients underwent isolated CABG and retrospectively followed to asses clinical outcomes of the two different revascularization techniques

SUMMARY:
Retrospective study of adult patients with multivessel disease undergoing isolated coronary artery bypass grafting (CABG) in three centers between January 1st, 2009, and December 31st, 2023. Patients were grouped according to the revascularization strategy (total arterial revascularization vs. multiarterial grafting). Primary outcome was a composite of major adverse cardiac and cerebrovascular events (MACCE).

ELIGIBILITY:
Inclusion Criteria:

* isolated CABG

Exclusion Criteria:

* single vessel CABG
* CABG with utilization of only one arterial graft

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients undergoing isolated CABG at Carmel medical center, Beilinson medical center and Soroka medical center at Israel
Sampling Method: Non-Probability Sample
Enrollment: 7878 (Actual)
Dates: Start 2009-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
MACCE | through study completion, a median of 101 months

SECONDARY OUTCOMES:
Mortality | through study completion, a median of 101 months
MI | through study completion, a median of 101 months
CVA | through study completion, a median of 101 months
repeat revascularization | through study completion, a median of 101 months